CLINICAL TRIAL: NCT01877746
Title: RANDOMIZED, MULTICENTRIC STUDY COMPARING THE EFFECT OF TWO REGIMENS OF COMBINED IMMUNOSUPPRESSIVE THERAPY IN THE TREATMENT OF INFLAMMATORY CARDIOMYOPATHY CZECH-ICIT (CZECH INFLAMMATORY CARDIOMYOPATHY IMMUNOSUPPRESSION TRIAL)
Brief Title: CZECH-ICIT (CZECH Inflammatory Cardiomyopathy Immunosuppression Trial)
Status: Unknown | Phase: Phase 3 | Type: Interventional
Last Known Status: Recruiting
Sponsor: St. Anne's University Hospital Brno, Czech Republic (Other)
Responsible Party: Principal Investigator, Jan Krejci, MD, Ph.D, MD, Ph.D, St. Anne's University Hospital Brno, Czech Republic
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: ICRC-ICIT-01
Record Dates: First submitted 2012-06-28; First posted 2013-06-14 (Estimated); Last update posted 2013-06-14 (Estimated); Status verified 2013-06

CONDITIONS: Inflammatory Cardiomyopathy
Keywords: ICM; myocarditis; cardiomyopathy; endomyocardial biopsy; immunosuppression
MeSH Terms: conditions — Myocarditis; Cardiomyopathies | interventions — Azathioprine

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (3):
- R1 - combined immunosuppressive therapy (Experimental): application of the combined immunosuppressive therapy in the first dosing regimen
  Interventions: Drug: Combination of prednisone and azathioprine
- R2 - combined immunosuppressive therapy (Experimental): application of the combined immunosuppressive therapy in the second dosing regimen
  Interventions: Drug: Combination of prednisone and azathioprine
- S - standard therapy (Other): only standard medical therapy of chronic heart failure without application of the combined immunosuppressive therapy
  Interventions: Other: No intervention

INTERVENTIONS:
Drug: Combination of prednisone and azathioprine — * Prednisone for a total of 90 days, with initial dose 1mg/kg/day p.o., given for 12 days and then tapered every 5 days for 5mg/day to the maintenance dose of 0.2mg/kg/day. The daily dose of Prednisone will be rounded to the nearest value divisible by 5.
  * Azathioprine for 100 days in total, with dose 1 mg/kg/day. The daily dose of Azathioprine will be rounded to the nearest value divisible by 25.
  Arms: R1 - combined immunosuppressive therapy
Drug: Combination of prednisone and azathioprine — * Prednisone for a total of 6 months, with initial dose 1mg/kg/day p.o. given for 4 weeks with a subsequent maintenance dose of 0,33 mg/kg/den. The daily dose of Prednisone will be rounded to the nearest value divisible by 5.
  * Azathioprine for 6 months in total, with dose 2mg/kg/day. The daily dose of Azathioprine will be rounded to the nearest value divisible by 25.
  Arms: R2 - combined immunosuppressive therapy
Other: No intervention — No intervention, only standard medical therapy
  Arms: S - standard therapy

SUMMARY:
The aim of this study is to compare the effect of combined immunosuppressive therapy given on the top standard medical therapy of chronic heart failure according to current guidelines with standard medical therapy of chronic heart failure alone in patients with infammatory cardiomyopathy (ICM).

Suitable subjects are characterized by EMB established presence of myocardial inflammation / negative polymerase chain reaction assay (PCR) findings of cardiotropic infectious agents and with varying duration of heart failure symptoms and left ventricular (LV) systolic dysfunction (phase A).

Further, to compare the effect of two regimens of combined immunosuppressive therapy in these patients with ICM (phase B).

ELIGIBILITY:
Inclusion Criteria:

1. Males and females aged 18 to 65 years at the time of signing the informed consent
2. Signing of the informed consent.
3. LV systolic dysfunction defined by ejection fraction less than/or equal 40% as assessed by echocardiography and symptoms of heart failure (minimum NYHA class II) lasting for at least 2 weeks at the time of randomization. This criterion also determines the inclusion of the study subjects in one of two substudies (CZECH-ICIT 1 or CZECH-ICIT 2).

   * LV systolic dysfunction (defined by ejection fraction less than/or equal 40%) and symptoms of heart failure (minimum NYHA class II) lasting 2 weeks to 6 months, with standard medical therapy of chronic heart failure given for at least 2 weeks - the subject fulfills criterion for inclusion in CZECH-ICIT 1 substudy
   * LV systolic dysfunction (defined by ejection fraction less than/or equal 40%) and symptoms of heart failure (minimum NYHA class II) lasting more than 6 months, with standard medical therapy of chronic heart failure given for at least 2 weeks - the subject fulfills criterion for inclusion in CZECH-ICIT 2 substudy
4. Positive immunohistochemistry finding of myocardial inflammation in endomyocardial biopsy (EMB). EMB must have been be performed no more than 6 weeks prior to the inclusion in the study. Positive immunohistochemistry EMB finding demonstrating myocardial inflammation is defined by the presence of at least 7/mm2 cluster of differentiation 3 (CD3) positive lymphocytes and/or at least 14 infiltrating leucocytes (LCA+ cells)/mm2 in the specimen.
5. The absence of infectious agent in EMB is defined by negative results of PCR testing of EMB specimens. PCR testing will be aimed to exclude the presence of enteroviruses (ECHO, coxsackie), adenoviruses, herpes viruses (herpes simplex virus (HSV-1), Epstein-Barr virus (EBV), cytomegalovirus (CMV), human herpes virus (HHV-6)), Borrelia burgdorferi and parvovirus B19. In the case of parvovirus B19, a negative PCR result will be considered when less than 500 viral copies/ug genomic DNA are detected. EMB must have been performed no more than 6 weeks prior to the inclusion in the study.
6. Negative blood pregnancy test in fertile females.
7. Usage of the effective method of contraception (hormonal or 2 barrier method of contraception)

Exclusion Criteria:

1. The presence of coronary artery disease, defined by angiographic findings of one or more coronary artery stenosis > 50%, history of previous myocardial infarction and/or percutaneous or surgical myocardial revascularization. Coronary angiography must not have been performed more than 2 years before randomization into the study.
2. Permanent pacemaker including cardiac resynchronization therapy.
3. The presence of uncontrolled, persistent supraventricular tachyarrhythmia, with ventricular rate > 120/min, lasting more than 1 week before EMB.
4. The presence of uncontrolled arterial hypertension, defined by blood pressure values > 180mmHg (for systolic pressure) and/or 110mmHg (for diastolic pressure) lasting more than 3 months.
5. The presence of at least moderately hemodynamically significant primary valvulopathy or congenital heart disease (apart from patent foramen ovale and non-significant atrial septal defect).
6. Previous heart valve surgery (replacement or reconstruction) or surgical correction of congenital heart disease. adu.
7. A history of cytostatic therapy or radiotherapy.
8. Alcoholism defined as ethanol intake >90 g/day.
9. The presence of uncontrolled endocrine of metabolic disorder.
10. Gravidity and lactation.
11. Known hypersensitivity to investigational drugs.
12. All contraindications of immunosuppressive therapy according to Summary of product characteristics (SmPC) of both investigational medicinal products: untreated systemic infection, poorly manageable diabetes mellitus, osteoporosis, florid gastric or duodenal ulcer, uncontrolled arterial hypertension, history of malignant disease with oncological treatment finished less than 5 years, proven immunodeficiency, renal of hepatic insufficiency (serum creatinine > 200 µmol/l; alanine aminotransferase (ALT) and/or aspartate aminotransferase (AST) activity greater than three times the standard), leukocytopenia (leucocytes less than 4 x 10 9/l), thrombocytopenia (platelets less than 100 x 10 9/l), anemia (hemoglobin concentration less than 100 g/l).

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 234 (Estimated)
Dates: Start 2013-01; Primary Completion 2015-09 (Estimated); Study Completion 2015-09 (Estimated)

PRIMARY OUTCOMES:
comparison of the change in LV ejection fraction | baseline and in 12 months after the initiation of immunosuppressive therapy

SECONDARY OUTCOMES:
comparison of the change of LV end-diastolic and end-systolic diameters | baseline and in 12 months after the initiation of immunosuppressive therapy
comparison of the change of New York Heart Association (NYHA) class | baseline and in 12 months after the initiation of immunosuppressive therapy
comparison of total mortality | baseline and in 12 months after the initiation of immunosuppressive therapy
comparison of the combined end-point | baseline and in 12 months after the initiation of immunosuppressive therapy
  combined end-point (death from cardiac reasons, heart transplantation, hospitalization for heart failure, successful resuscitation for cardiac arrest and adequate implantable cardioverter-defibrillator (ICD) shock for ventricular tachycardia or fibrillation
comparison of the change in the number of infiltrating inflammatory cells in EMB | baseline and in 12 months after the initiation of immunosuppressive therapy

CONTACTS AND LOCATIONS:
Overall Officials: Jan Krejci, MD, Ph.D, Principal Investigator — employee; Tomas Palecek, Assoc. prof., Principal Investigator — without affiliation
Locations (2):
- Czechia (2):
  - St. Anne's University Hospital Brno, Brno
  - General University hospital in Prague, Prague

REFERENCES:
- [Background] Wojnicz R, Nowalany-Kozielska E, Wojciechowska C, Glanowska G, Wilczewski P, Niklewski T, Zembala M, Polonski L, Rozek MM, Wodniecki J. Randomized, placebo-controlled study for immunosuppressive treatment of inflammatory dilated cardiomyopathy: two-year follow-up results. Circulation. 2001 Jul 3;104(1):39-45. doi: 10.1161/01.cir.104.1.39. PMID 11435335
- [Background] Frustaci A, Russo MA, Chimenti C. Randomized study on the efficacy of immunosuppressive therapy in patients with virus-negative inflammatory cardiomyopathy: the TIMIC study. Eur Heart J. 2009 Aug;30(16):1995-2002. doi: 10.1093/eurheartj/ehp249. Epub 2009 Jun 25. PMID 19556262